CLINICAL TRIAL: NCT07115914
Title: Prospective Evaluation of PSMA PET Imaging in Surveillance Post-Focal Therapy for Prostate Cancer (PSMA-FT Surveillance Study)
Brief Title: Monitoring Patient Prostate Health Post Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Blue Earth Diagnositcs (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 24-2132
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer (Adenocarcinoma); Prostate Cancer (Diagnosis); Prostate Cancer Metastatic Disease
Keywords: focal therapy; prostate cancer; prostate cancer patient
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): All people enrolled in this study will participate in the same study arm and will receive the same study interventions.
  Interventions: Radiation: PSMA PET/CT scan

INTERVENTIONS:
Radiation: PSMA PET/CT scan — A PSMA PET scan, or prostate-specific membrane antigen positron emission tomography scan, is an imaging test that scans and takes pictures of the prostate. PSMA scans use a specialized radioactive imaging dye that sticks to the proteins that are typically found in prostate cancer cells. This imaging dye helps locate areas of prostate cancer anywhere in the body, both inside and outside prostate.

SUMMARY:
This study is about adding PSMA PET (Prostate Specific Membrane Antigen- Positron Emission Tomography) to routine magnetic resonance imaging (MRI) scans to help detect prostate cancer recurrence in men who have undergone focal therapy for prostate cancer. PSMA PET and multiparametric (mpMRI are both imaging tests that help detect prostate cancer in the body.

A PSMA PET scan, or prostate-specific membrane antigen positron emission tomography scan, is an imaging test that scans and takes pictures of the prostate. PSMA scans use a specialized radioactive imaging dye that sticks to the proteins that are typically found in prostate cancer cells. This imaging dye helps locate areas of prostate cancer anywhere in the body, both inside and outside prostate.

An mpMRI, or a multiparametric (mp) MRI scan, is also an imaging test that scans and takes detailed pictures of the prostate. Unlike regular MRIs, an mpMRI produces a more detailed image of the prostate. Similar to PET scans, mpMRI scans also use an imaging dye that helps the pictures of the prostate appear clearer on scans.

This study will be funded by Blue Earth Diagnostics, a molecular imaging company based in England.

DETAILED DESCRIPTION:
People who agree to join the study will be asked to attend study visits for about 12 months after focal therapy. Focal therapy will not be given as part of research in this study. Study participants will receive focal therapy, a follow up MRI and prostate biopsy as part of regular clinical care for their cancer. This research study will add an additional PSMA PET to follow up after focal therapy.

Study participants will also be asked to:

* Give blood, urine and tissue samples for research purposes. The decision to give tissue samples is optional and not required for participation in study.
* Fill out quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be male (assigned male at birth) and 18 years or older.
2. Subjects must demonstrate the ability to understand and provide written informed consent.
3. Subjects must have histologically confirmed prostate cancer ( PCa) Note: Recruitment will be limited to a maximum of 50% of subjects with favorable intermediate-risk prostate cancer (PCa) Note: The histopathologic diagnosis must be obtained via "Prostate Biopsy (PB)", which for the purposes of the present study, is defined as both a systematic 12-core sextant random prostate biopsy and a targeted prostate biopsy. The targeted prostate biopsy can be performed via in-bore multiparemetric (mp) magnetic resonance imaging (MRI) prostate biopsy, cognitive mpMRI/ultrasound fusion prostate biopsy or software mpMRI/ultrasound fusion prostate biopsy. This "PB" must not be obtained greater than 1 year from the date of consent.
4. Subjects must have chosen to get focal therapy (partial gland ablation) for the treatment of prostate cancer and must be scheduled for partial gland ablation/focal therapy with any energy modality within 6 months following informed consent.
5. Subjects must have confirmed non-metastatic PCa following SOC screening for patients with unfavorable intermediate-risk and high risk PCa, a combination of computed tomography imaging of the abdomen and pelvis (CTAP) and technetium-99-mDP nuclear medicine bone scan (BS) and/or PSMA-PET imaging prior to enrollment. The imaging studies should be obtained within 6-months of enrollment.
6. Subjects must be designated as Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 or Karnofsky Performance Status Scale Score ≥ 60%, (see Appendix A).
7. Subjects must be fit to undergo general anesthesia and the FT surgical procedure, which includes adequate visualization of the prostate gland on transrectal ultrasound imaging, access to the urethra, perineum and rectum, as well as be tolerant of lithotomy positioning in the opinion of the treating investigator or the operating surgeon(s) if not the same as the treating investigator.

Exclusion Criteria:

1. Subject had prior or current PCa therapies, such as biologic, chemotherapy, hormone therapy, radiotherapy or surgery for PCa within last 12 months. Subjects who received radiation and/or androgen deprivation therapy for prostate cancer more than 12 months prior to diagnosis of recurrent prostate cancer will be eligible for the trial.
2. Subjects with locally advanced, nodal or metastatic prostate cancer.
3. Subjects who are unfit for pelvic mpMRI scanning (e.g., severe claustrophobia), permanent cardiac pacemaker, metallic implants that are likely to contribute to significant image artifacts, allergy or contraindication to gadolinium contrast agent.
4. If the subject has an uncontrolled or major debilitating inter-current illness.
5. Judgment by the treating investigator or PI that the subject is unsuitable to participate in the study and the subject is unlikely to comply with study procedures, restrictions, and requirements.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer
Enrollment: 62 (Estimated)
Dates: Start 2027-08-01 (Estimated); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
PSMA-PET combined with mpMRI to Assess Prostate Cancer Risk | 1 year
  PSMA-PET combined with mpMRI to differentiate a patient's risk for prostate cancer as assessed by Gleason Scores and radiology/clinical notes.

SECONDARY OUTCOMES:
PSMA-PET combined with MpMRI to Select Patients for Partial Gland Ablation | 1 year
  PSMA-PET in combination with MpMRI imaging for selecting patients for partial gland ablation as assessed by clinical investigator.
PSMA-PET combined with PSA to Diagnose Cancer Recurrence After Partial Gland Ablation | 1 year
  PSMA-PET in combination with PSA for diagnosing clinically significant cancer recurrence/residual disease after partial gland ablation.

CONTACTS AND LOCATIONS:
Overall Officials: Abhinav Sidana, MD, Principal Investigator — University of Chicago

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF